CLINICAL TRIAL: NCT02653079
Title: Immunophenotyping From Blood of Patients Suffering From Chronic Degenerating Joint Diseases and Receiving Local Low Dose Radiation Therapy (LDRT)
Brief Title: Immunophenotyping From Blood of Patients Suffering From Chronic Degenerating Joint Diseases and Receiving LDRT
Acronym: IMMO-LDRT01
Status: Recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: IMMO-LDRT01
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Chronic Inflammatory Disorder
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, Blood cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Cohort: Blood draw and Questionaire from patients suffering from chronic inflammatory diseases of the joints, namely painful shoulder syndrome (periarthritis humeroscapularis), painful elbow syndrome (Epicondylopathia humeri), benign achillodynia, and benign calcaneodynia, Arthrosis (finger- and Rhizarthrosis, Gonarthrosis, Anklearthrosis), and Arthritis with an planned local low dose radiation therapy (LDRT) at the Department of Radiation Oncology, Universitätsklinikum Erlangen.
  Interventions: Other: Blood Draw and Questionaire

INTERVENTIONS:
Other: Blood Draw and Questionaire — The study is observational. The treatment-plan of the underlying disease remained unchanged. Blood draw from patients at several time points during and after low dose radiation therapy.

SUMMARY:
Patients suffering from chronic degenerating diseases are often treated by a plethora of NSAIDs, DMARDs, Biologicals, as well as combinations of these therapeutics. However, many patients are refractory to this treatment and suffer from chronic pain over years, leading to a worsening of the quality of live. The mobilization of these patients is one main goal in the therapy of these chronic and inflammatory diseases. Low dose radiation therapy (LDRT) is applied since more than one century for the local treatment of chronic degenerating joint diseases. The success of the treatment was described by many retrospective as well as pattern of care studies, respectively.

Local (only at the painful joint) low dose irradiation of the chronic patients results in most patients in a significantly reduced pain, not only direct after the therapy, but also lasting for more than 12 month in many cases. The patients experience enhanced mobility and increased quality of life. The molecular and cellular processes leading to the pain reduction are just fragmentarily analyzed. Our group revealed that macrophages are key players in radiation-induced immune modulation. Inflammatory macrophages exposed to low doses of radiation showed a reduced inflammatory capacity and attenuated an inflammatory microenvironment. Besides macrophages further immune cells are most likely involved in reduction of inflammation following LD-RT, as in vitro already shown for neutrophils.

The IMMO-LDRT01 study aims for the first time to analyze in detail the immune status of patients suffering from inflammatory, chronic joint diseases before, during and after LD-RT in a longitudinal manner. The multi-color flow cytometry-based assay will allow determining over 30 immune cell subsets and additionally their activation status. Further, biodosimetry will be performed with the whole-blood samples to get hints about dose that the immune cells are exposed to. This will be performed with national and international co-operation partners.

The IMMO-LDRT01 study is a prospective and observational study not influencing the standard therapeutic scheme and will provide hints how the LDRT affects besides local cells in the irradiated area also the systemic inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering and diagnosed for:
* painful shoulder syndrome (periarthritis humeroscapularis)
* painful elbow syndrome (Epicondylopathia humeri)
* benign achillodynia
* benign calcaneodynia
* arthosis (finger- , rhiz-, gon-, and anklearthrosis
* arthritis (gon- and anklearthrosis)
* Planned local low dose radiation therapy (LDRT) at the Department of Radiation Oncology, Universitätsklinikum Erlangen.
* Age at least 18 years

Exclusion Criteria:

* patients who are suffering or had suffered from any malignant diseases
* fertile patients who refuse effective contraception during study treatment
* persistent drug and/or alcohol abuse
* patients not able or willing to behave according to study protocol
* patients in care
* patients that are not able to speak German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from chronic inflammatory diseases of the joints, namely painful shoulder syndrome (periarthritis humeroscapularis), painful elbow syndrome (Epicondylopathia humeri), benign achillodynia, benign calcaneodynia, arthosis (finger- , rhiz-, gon-, and anklearthrosis, and arthritis (gon- and anklearthrosis).
  Patients were attributed to our clinic and the study protocol was explained in detail. The patients have to give their informed consent before starting with the LDRT. The treatment-plan of the underlying disease remained unchanged. This treatment scheme is conducted with 2 irradiations within 7 days for total treatment duration of 3 weeks. The single dose is 0.5 Gy and the complete dose of one round of LDRT is 3 Gy.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-06; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change of circulating immune cells of treated patients by deep immunophenotyping. | up to 3 month after completion of RT
  Immunophenotyping of the patients: Detection of about 30 distinct immune sell (sub)types together with their activation markers. The analyses are conducted at time points before (day 0) and after low dose radiation therapy (day 21): before LDRT (day 0), end of first round of LDRT (last day of LDRT, usually at 3 Gy), and 3 month (day 111) after completed RT. This scheme is repeated if patient receives additional round of LDRT for relapse treatment.

SECONDARY OUTCOMES:
Change of joint pain intensity of the treated patients. | up to 9 month after completion of RT
  Analysis of the pain by VAS (visaul Analog Scale; 0 - lowest pain intensity, 10 highest pain intensity) at time points before and after low dose radiation therapy: before LDRT (day 0), end of first round of LDRT (last day of LDRT, usually at 3 Gy), and 3 month (day 111) after completed RT. This scheme is repeated if patient receives additional round of LDRT for relapse treatment.
Change of functional capacity in daily life of the treated patients | up to 9 month after completion of RT
  Analysis of the functional capacity in daily life by FFbH-R (Funktionsfragebogen Hannover, 100% normal to 10 % nearly complete restricted) questionnaire at time points before and after low dose radiation therapy: before LDRT (day 0), end of first round of LDRT (last day of LDRT, usually at 3 Gy), and 3 month (day 111) after completed RT. This scheme is repeated if patient receives additional round of LDRT for relapse treatment.
Change of health-related quality of life | up to 9 month after completion of RT
  Analysis of the health-related quality of life by EQ5DL (health index value) questionnaire at time points before and after low dose radiation therapy: before LDRT (day 0), end of first round of LDRT (last day of LDRT, usually at 3 Gy), and 3 month (day 111) after completed RT. This scheme is repeated if patient receives additional round of LDRT for relapse treatment.
description of pain quality | up to 9 month after completion of RT
  Analysis of the pain by descriptive questionnaire at time points before and after low dose radiation therapy: before LDRT (day 0), end of first round of LDRT (last day of LDRT, usually at 3 Gy), and 3 month (day 111) after completed RT. This scheme is repeated if patient receives additional round of LDRT for relapse treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver J Ott, MD, Principal Investigator — Department of Radiation Oncology, Universitätsklinikum Erlangen, Friedrich-Alexander-Universität Erlangen-Nürnberg; Udo S Gaipl, PhD, Principal Investigator — Department of Radiation Oncology, Universitätsklinikum Erlangen, Friedrich-Alexander-Universität Erlangen-Nürnberg
Locations (1):
- Department of Radiation Oncology, Universitätsklinikum Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Donaubauer AJ, Becker I, Weissmann T, Frohlich BM, Munoz LE, Gryc T, Denzler M, Ott OJ, Fietkau R, Gaipl US, Frey B. Low Dose Radiation Therapy Induces Long-Lasting Reduction of Pain and Immune Modulations in the Peripheral Blood - Interim Analysis of the IMMO-LDRT01 Trial. Front Immunol. 2021 Oct 12;12:740742. doi: 10.3389/fimmu.2021.740742. eCollection 2021. PMID 34712229